CLINICAL TRIAL: NCT04278209
Title: Measurement of Glycogen Replenishment in Children After an Overnight Fast
Brief Title: Glycogen Metabolism in Children
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Société des Produits Nestlé (SPN) (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: 1906NRC
Record Dates: First submitted 2020-02-18; First posted 2020-02-20 (Actual); Last update posted 2022-01-26 (Actual); Status verified 2022-01

CONDITIONS: Healthy
MeSH Terms: interventions — Water

STUDY DESIGN:
Intervention Model Description: Randomized, controlled, balanced incomplete crossover design
Masking Description: Open Label
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (6):
- Breakfast 1 - Breakfast 2 (Experimental): Participants will receive Breakfast 1 then Breakfast 2.
  Interventions: Other: Breakfast 1; Other: Breakfast 2
- Breakfast 1 - water (Experimental): Participants will receive Breakfast 1, then water.
  Interventions: Other: Breakfast 1; Other: Water
- Breakfast 2 - water (Experimental): Participants will receive Breakfast 2, then water.
  Interventions: Other: Breakfast 2; Other: Water
- Breakfast 2 - Breakfast 1 (Experimental): Participants will receive 2 servings, then 1 serving of the study product.
  Interventions: Other: Breakfast 1; Other: Breakfast 2
- Water - Breakfast 1 (Experimental): Participants will receive water, then Breakfast 1.
  Interventions: Other: Breakfast 1; Other: Water
- Water - Breakfast 2 (Experimental): Participants will receive water, then Breakfast 2.
  Interventions: Other: Breakfast 2; Other: Water

INTERVENTIONS:
Other: Breakfast 1 — Participant will receive Breakfast 1
  Arms: Breakfast 1 - Breakfast 2; Breakfast 1 - water; Breakfast 2 - Breakfast 1; Water - Breakfast 1
Other: Breakfast 2 — Participant will receive Breakfast 2
  Arms: Breakfast 1 - Breakfast 2; Breakfast 2 - Breakfast 1; Breakfast 2 - water; Water - Breakfast 2
Other: Water — Participant will receive water
  Arms: Breakfast 1 - water; Breakfast 2 - water; Water - Breakfast 1; Water - Breakfast 2

SUMMARY:
It is not fully understood in children how much of hepatic and muscle glycogen is used during a night and how they are replenished after a breakfast. This study aims to analyze the glycogen metabolism before and after an overnight sleep as well as after a breakfast in children between 8 and 12 years old.

DETAILED DESCRIPTION:
The aim of the study is to investigate if liver and muscle glycogen stores are depleted in children after overnight fasting and to what extend the stores are replenished with the intake of small breakfast.

The study is a balanced incomplete crossover design. Participants (children between 8 and 12 years old) have to be two periods of two days in the study. They will be randomized in 6 arms, receiving either water, 1 serving of a small breakfast (Breakfast 1) or 2 servings of the small breakfast (Breakfast 2).

An Interim Analysis after 9 completed subjects will be performed in order to calculate the total number of subjects needed to adequately power the Primary Endpoint.

ELIGIBILITY:
Inclusion Criteria:

1. Healthy girls and boys between 8 and 12 years of age
2. Clinically healthy body weight (5 to 85th rounded percentile from UK)
3. In good health as determined by health screening questionnaires
4. English proficiency as per investigator judgment
5. Informed consent signed by parent(s), or legal representative if applicable and signed child assent according to local legislation

Exclusion Criteria:

1. Girls having menstruations
2. Any type of self-reported food allergies
3. Lactose intolerance
4. Claustrophobic
5. Diagnosis of Diabetes Mellitus
6. Diagnosed acute or chronic medical conditions that could impact study outcomes (asthma)
7. Ongoing diseases or intake of any prescribed or over the counter drugs
8. Participants or participants' parent(s) or legal representative who are not willing and not able to comply with scheduled visits and the requirements of the study protocol (including a consumption of 200 ml study drink)
9. Currently participating or having participated in another clinical trial within 12 weeks prior to trial start.

Ages: 8 Years to 12 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 24 (Actual)
Dates: Start 2020-01-23 (Actual); Primary Completion 2021-11-30 (Actual); Study Completion 2021-11-30 (Actual)

PRIMARY OUTCOMES:
Incremental/decremental AUC0-240 of the concentration/time curve of hepatic glycogen | 4 hours
  To determine the effects of 1 and 2 servings of a small breakfast on hepatic glycogen stores; measured by NMR

SECONDARY OUTCOMES:
Change of hepatic glycogen content over an overnight fast | 12 hours
  Change of hepatic glycogen content over an overnight fast
Change of muscle glycogen content over an overnight fast | 12 hours
  Change of muscle glycogen content over an overnight fast
Incremental/decremental AUC0-240 of the concentration/time curve of muscle glycogen | 4 hours
  To determine the effects of 1 and 2 servings of a small breakfast on muscle glycogen stores; measured by NMR

CONTACTS AND LOCATIONS:
Overall Officials: Liz Simpson, PhD, Principal Investigator — University of Nottingham Medical School
Locations (1):
- University of Nottingham Medical School, Nottingham, United Kingdom

REFERENCES:
- [Derived] Horstman AM, Bawden SJ, Spicer A, Darwish N, Goyer A, Egli L, Rupp N, Minehira K, Gowland P, Breuille D, Macdonald IA, Simpson EJ. Liver glycogen stores via 13C magnetic resonance spectroscopy in healthy children: randomized, controlled study. Am J Clin Nutr. 2023 Apr;117(4):709-716. doi: 10.1016/j.ajcnut.2023.01.014. Epub 2023 Jan 20. PMID 36797201